CLINICAL TRIAL: NCT02400255
Title: A Phase II Study of Crenolanib Besylate Maintenance Following Allogeneic Stem Cell Transplantation in Patients With FLT3-positive Acute Myeloid Leukemia
Brief Title: Crenolanib Maintenance Following Allogeneic Stem Cell Transplantation in FLT3-positive Acute Myeloid Leukemia Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Arog Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ARO-009
Record Dates: First submitted 2015-03-18; First posted 2015-03-27 (Estimated); Results first posted 2023-12-18 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2023-12

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cohort A (Experimental): Cohort A will include patients who underwent allogeneic hematopoietic stem cell transplantation (HSCT) while in first or second complete remission with count recovery. Crenolanib besylate maintenance therapy will start at the earliest time no sooner than 42 days but no later than 90 days after allogeneic HSCT.
  Interventions: Drug: Crenolanib besylate
- Cohort B (Experimental): Cohort B will include patients who underwent HSCT with incomplete count recovery although they had ≤%10 bone marrow blasts at the time of HSCT. Crenolanib besylate maintenance therapy will start at the earliest time no sooner than 42 days but no later than 90 days after allogeneic HSCT.
  Interventions: Drug: Crenolanib besylate

INTERVENTIONS:
Drug: Crenolanib besylate
  Other Names: CP-868,596-26

SUMMARY:
This is a single-arm, Phase II study of crenolanib as maintenance in AML patients with FLT3 mutations who have achieved complete remission (CR) after allogeneic stem cell transplantation. Oral crenolanib will be administered daily post-transplant for up to two years.

DETAILED DESCRIPTION:
There are two patient subgroups: 1) those who were in complete remission (CR) at the time of transplant, and 2) those who were not in complete remission (NCR) at the time of transplant. Start of crenolanib therapy at 100 mg TID is intended at the earliest time no sooner than 42 days but no later than 90 days after allogeneic stem cell transplantation. Patients may take crenolanib continuously for up to 728 days or until one of the criteria for study discontinuation is fulfilled.

ELIGIBILITY:
Inclusion Criteria:

1. History of AML according to World Health Organization (WHO) classification
2. First allogeneic hematopoietic stem cell transplantation (HSCT) using myeloablative conditioning (MAC), non-myeloablative (NMA), or reduced-intensity conditioning (RIC) preparative regimens.
3. FLT3-ITD or FLT3-D835 positive disease at any time during disease course.
4. Hematopoietic stem cell source is either with peripheral blood, bone marrow or cord blood.
5. Donor source is matched related, unrelated, haploidentical donor or cord blood.
6. At the time of allogeneic HSCT:

   1. No more than 1 antigen mismatch at HLA-A, -B, -C, -DRB1 or -DQB1 locus for unrelated donor with peripheral blood and bone marrow as the hematopoietic stem cell source; and
   2. Bone marrow blast ≤ 10%
7. No sooner than 42 days but no later than 90 days after allogeneic HSCT.
8. Post-transplant bone marrow blast count ≤ 5% confirmed within 21 days (+4 days) prior to starting study therapy
9. Evidence of donor engraftment as defined by institutional standard T cell chimerism > 50%.
10. Adequate engraftment within 7 days prior to starting study therapy: ANC ≥ 1.0 x 10^9/L without daily use of myeloid growth factor; and platelet ≥ 25 x 10^9/L without platelet transfusion within 1 week
11. Non-hematological toxicities ≤ Grade 2
12. Serum creatinine ≤ 1.5 × ULN OR creatinine clearance ≥ 50mL/min/1.73 m2 for subjects with creatinine levels above institutional normal
13. Adequate liver function with serum AST, ALT and bilirubin within the normal range at the time of crenolanib commencement
14. Acute graft-versus-host disease (GVHD) ≤ Grade 1, either no signs of chronic GVHD or mild chronic GVHD graded as limited disease
15. Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
16. Age ≥ 18 years with the capacity to give written informed consent
17. Non-pregnant and non-nursing women of childbearing potential must have a negative serum or urine pregnancy test ("Women of childbearing potential" is defined as a sexually active mature woman who has not undergone a hysterectomy or who has had menses at any time in the preceding 24 consecutive months)
18. Women of childbearing potential and men must agree to use adequate contraception prior to study entry, for the duration of study participation and for 90 days following completion of therapy

Exclusion Criteria:

1. Bone marrow blast >5% within 21 days (+4 days) of start of study drug
2. Active GVHD grade ≥ 2
3. Concurrent use of corticosteroids equivalent of prednisone at a dose > 0.5 mg/kg
4. Active and/or untreated central nervous system (CNS) leukemia
5. Concomitant therapies for treatment or control of leukemia.
6. Use of any of the following after transplantation and prior to starting study therapy:

   1. Chemotherapeutic agents for therapy of AML (note that prophylactic use of these agents is allowed in this study, e.g., methotrexate for GVHD)
   2. Investigational agents/therapies
   3. Azacitidine, decitabine or other demethylating agents
   4. Lenalidomide, thalidomide and pomalidomide
7. Uncontrolled infection
8. Known positive for human immunodeficiency virus (HIV); active hepatitis B (HBV) or hepatitis C (HCV) infection
9. Significant cardiac disease (New York Heart Association classes III or IV) or unstable angina despite medication
10. Pregnant or breast-feeding
11. Major surgery within 4 weeks of starting study drug
12. Receipt of investigational agents within 5 half-lives of last dose of investigational agent
13. Prior treatment with crenolanib with progression on treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2022-05 (Actual); Study Completion 2022-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Champlin, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Patients in Complete Remission 1 (CR1): Subjects who underwent allogeneic hematopoietic stem cell transplantation (HSCT) while in first complete remission with count recovery received crenolanib besylate maintenance therapy. Maintenance was started at the earliest time no sooner than 45 days but no later than 90 days after allogeneic HSCT.
- Patients in Complete Remission 2 (CR2): Subjects who underwent allogeneic hematopoietic stem cell transplantation (HSCT) while in second complete remission with count recovery received crenolanib besylate maintenance therapy. Maintenance was started at the earliest time no sooner than 45 days but no later than 90 days after allogeneic HSCT.
- Patients in Complete Remission 3 (CR3): Subjects who underwent allogeneic hematopoietic stem cell transplantation (HSCT) while in third complete remission with count recovery received crenolanib besylate maintenance therapy. Maintenance was started at the earliest time no sooner than 45 days but no later than 90 days after allogeneic HSCT.
- Residual Disease: Subjects who underwent allogeneic hematopoietic stem cell transplantation (HSCT) with incomplete count recovery and bone marrow blasts ≤%10 received crenolanib besylate maintenance therapy. Maintenance was started at the earliest time no sooner than 45 days but no later than 90 days after allogeneic HSCT.
Period: Overall Study
Arm/Group | Patients in Complete Remission 1 (CR1) | Patients in Complete Remission 2 (CR2) | Patients in Complete Remission 3 (CR3) | Residual Disease
Started | 22 | 5 | 1 | 2
Completed | 5 | 1 | 0 | 0
Not Completed | 17 | 4 | 1 | 2
Not completed — Relapse | 4 | 1 | 1 | 2
Not completed — Adverse Event | 6 | 3 | 0 | 0
Not completed — Physician Decision | 6 | 0 | 0 | 0
Not completed — Loss of insurance | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Patients in Complete Remission 1 (CR1) | Patients in Complete Remission 2 (CR2) | Patients in Complete Remission 3 (CR3) | Residual Disease | Total
Number analyzed (Participants) | 22 | 5 | 1 | 2 | 30
Age, Continuous [Median (Full Range); unit: years] | 54.5 [24 to 69] | 53 [47 to 71] | 37 [37 to 37] | 61 [48 to 74] | 53.5 [24 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 1 | 0 | 2 | 14
  Male | 11 | 4 | 1 | 0 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 0 | 0 | 4
  Not Hispanic or Latino | 18 | 2 | 1 | 2 | 23
  Unknown or Not Reported | 2 | 1 | 0 | 0 | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 1 | 0 | 0 | 0 | 1
  Asian | 2 | 0 | 0 | 0 | 2
  White | 14 | 5 | 1 | 2 | 22
  Other | 5 | 0 | 0 | 0 | 5
FLT3 Mutations [Count of Participants; unit: Participants] — Mutations in the gene encoding the trans-membrane tyrosine kinase FLT3. The type of FLT3 mutation detected by bone marrow assessment at diagnosis was collected. Subjects had either internal tandem duplications (ITD) in the juxtamembrane domain, point mutations or deletions in the tyrosine kinase domain (TKD) or both ITD and TKD mutations together.
  Participants
    ITD only | 18 | 4 | 1 | 1 | 24
    TKD only | 3 | 1 | 0 | 1 | 5
    ITD and TKD | 1 | 0 | 0 | 0 | 1
AML diagnosis [Count of Participants; unit: Participants] — Whether or not subjects had a prior history of antecedent hematological disease. Subjects with de novo AML do not have a history of antecedent hematological disease, while subjects with secondary AML do.
  Participants
    De novo AML | 20 | 4 | 1 | 2 | 27
    Secondary AML (CMML or MDS) | 2 | 1 | 0 | 0 | 3
Conditioning regimen [Count of Participants; unit: Participants] — The type of chemotherapy regimen the subjects received prior to hematopoietic stem cell transplant. Reduced intensity conditioning refers to a regimen that uses less chemotherapy and/or radiation than the standard myeloablative regimen.
  Participants
    Myeloablative | 16 | 3 | 1 | 2 | 22
    Reduced intensity | 6 | 2 | 0 | 0 | 8
Donor type [Count of Participants; unit: Participants] — The type of donor cells used in the subject's hematopoietic stem cell transplant. Matched related stem cells refer to donor cells harvested from a relative with matching human leukocyte antigen. Matched unrelated stem cells refer to donor cells harvested from an unrelated individual with matching human leukocyte antigen. Haploidentical stem cells refer to donor cells harvested from half human leukocyte antigen matched relatives.
  Participants
    Matched related | 9 | 2 | 1 | 1 | 13
    Matched unrelated | 10 | 3 | 0 | 1 | 14
    Haploidentical | 3 | 0 | 0 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Who Relapsed
Description: Patients who relapsed during or after crenolanib maintenance therapy were categorized as those who received <28 days of maintenance and those who received >28 days of maintenance.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Groups:
- All Subjects: Subjects who underwent allogeneic hematopoietic stem cell transplantation (HSCT) while either in first, second or third complete remission with count recovery or with incomplete count recovery and bone marrow blasts ≤%10 received crenolanib besylate maintenance therapy. Maintenance was started at the earliest time no sooner than 45 days but no later than 90 days after allogeneic HSCT.
Arm/Group | All Subjects | Patients in Complete Remission 1 (CR1) | Patients in Complete Remission 2 (CR2) | Patients in Complete Remission 3 (CR3) | Residual Disease
Number analyzed (Participants) | 30 | 22 | 5 | 1 | 2
Participants
  Early relapses within the first 28 days of treatment | 5 | 2 | 0 | 1 | 2
  Relapses after the first 28 days of treatment | 4 | 3 | 1 | 0 | 0

ADVERSE EVENTS:
Time Frame: 2 years
Description: Safety data was presented in a comprehensive manner since no formal arms existed as part of the study; patients were only categorized this way during post-study data analyses to determine if there was a potential relationship between their disease status prior to transplant and their response to maintenance therapy.
Groups:
- All Patients: Subjects who underwent allogeneic hematopoietic stem cell transplantation (HSCT) while either in first, second or third complete remission with count recovery or with incomplete count recovery and bone marrow blasts ≤%10 received crenolanib besylate maintenance therapy. Maintenance was started at the earliest time no sooner than 45 days but no later than 90 days after allogeneic HSCT.
Arm/Group | All Patients
All-Cause Mortality (participants affected / at risk) | 9/30
Serious Adverse Events (participants affected / at risk) | 14/30
Other Adverse Events (participants affected / at risk) | 30/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Patients (N=30)
Anemia (Blood and lymphatic system disorders) | 3
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Pain (General disorders) | 1
Pyrexia (General disorders) | 3
Biliary dyskinesia (Hepatobiliary disorders) | 1
Infection (Infections and infestations) | 3
Influenza (Infections and infestations) | 1
Lung infection (Infections and infestations) | 2
Pneumonia (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Alanine aminotransferase increased (Investigations) | 1
Blood creatinine increased (General disorders) | 1
Platelet count decreased (Investigations) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 2
Cerebrovascular accident (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Presyncope (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 2
Mental status changes (Psychiatric disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 3
Haematuria (Renal and urinary disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Hypotension (Vascular disorders) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | All Patients (N=30)
Anemia (Blood and lymphatic system disorders) | 6
Febrile neutropenia (Blood and lymphatic system disorders) | 2
Sinus bradycardia (Cardiac disorders) | 2
Periorbital oedema (Eye disorders) | 3
Abdominal pain (Gastrointestinal disorders) | 3
Constipation (Gastrointestinal disorders) | 4
Diarrhoea (Gastrointestinal disorders) | 14
Dyspepsia (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 18
Vomiting (Gastrointestinal disorders) | 14
Face oedema (General disorders) | 2
Fatigue (General disorders) | 5
Localised oedema (General disorders) | 3
Oedema peripheral (General disorders) | 5
Pyrexia (General disorders) | 5
Graft versus host disease in gastrointestinal tract (Immune system disorders) | 2
Graft versus host disease in skin (Immune system disorders) | 3
Herpes zoster (Infections and infestations) | 3
Infection (Infections and infestations) | 3
Influenza (Infections and infestations) | 2
Lung infection (Infections and infestations) | 2
Pneumonia (Infections and infestations) | 4
Sinusitis (Infections and infestations) | 3
Staphylococcal infection (Infections and infestations) | 2
Upper respiratory tract infection (Infections and infestations) | 7
Urinary tract infection (Infections and infestations) | 3
Urinary tract infection enterococcal (Infections and infestations) | 2
Alanine aminotransferase increased (Investigations) | 6
Aspartate aminotransferase increased (Investigations) | 3
Blood alkaline phosphatase increased (Investigations) | 4
Blood creatinine increased (Investigations) | 5
Neutrophil count decreased (Investigations) | 2
Platelet count decreased (Investigations) | 12
Decreased appetite (Metabolism and nutrition disorders) | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 4
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2
Hypokalaemia (Metabolism and nutrition disorders) | 2
Hyponatraemia (Metabolism and nutrition disorders) | 2
Dizziness (Nervous system disorders) | 3
Paraesthesia (Nervous system disorders) | 2
Syncope (Nervous system disorders) | 2
Acute kidney injury (Renal and urinary disorders) | 3
Haematuria (Renal and urinary disorders) | 2
Rash (Skin and subcutaneous tissue disorders) | 3
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 6
Swelling face (Skin and subcutaneous tissue disorders) | 2
Hypotension (Vascular disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-06): https://cdn.clinicaltrials.gov/large-docs/55/NCT02400255/Prot_SAP_000.pdf